CLINICAL TRIAL: NCT03397238
Title: Myeloid Cell Reprogramming in the Context of Radioiodine Therapy in Patients With Non-Medullary Thyroid Carcinoma
Brief Title: Myeloid Cell Reprogramming in Thyroid Carcinoma
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL62671.091.17; 2017-3628 (Other: CMO Arnhem-Nijmegen)
Record Dates: First submitted 2017-12-18; First posted 2018-01-11 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2020-11

CONDITIONS: Thyroid Cancer
Keywords: myeloid cell; reprogramming; monocyte; tumor-associated macrophage
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Non-metastatic TC: blood withdrawal, bone marrow aspiration
- Metastatic TC: blood withdrawal, bone marrow aspiration
- MNG surgery: blood withdrawal, bone marrow aspiration
- MNG RAI treatment: blood withdrawal
- Healthy volunteers: blood withdrawal

SUMMARY:
This study investigates the reprogramming of myeloid cells in patients with thyroid carcinoma. The investigators hypothesize that tumor-derived factors change the function of myeloid cells (peripheral blood and bone marrow-derived) in such a way that these immune cells promote tumor growth rather than combat the tumor.

DETAILED DESCRIPTION:
Description of the problem:

Non-medullary thyroid carcinoma (TC) is the most common endocrine malignancy and its incidence is one of the most rapidly increasing among the cancer types. For many patients with advanced and poorly differentiated tumors, treatment options are limited and the prognosis of advanced stage metastatic disease remains poor.

Envisioned solution/research direction:

To improve the patients outcome and identify novel therapeutic targets, one needs a 'systems understanding' of the pathophysiology of tumors, particularly the complex interaction of the malignant cells with other cell types in the tumor en the tumor environment (TME), especially immune cells. Tumor-associated macrophages (TAMs), the most dominant myeloid population in aggressive thyroid tumors, exhibit a distorted phenotype functioning predominantly as tumor enhancer. Despite the progress in understanding the importance of TAMs, the in-depth characterization of different TAMs populations is lacking and the mechanisms governing the functional polarization of TAMs are largely unknown. Understanding the interplay between TAMs and tumor cells represents a crucial step towards development of additional therapeutic strategies in cancer.

Hypothesis:

1. We first propose that in advanced TC, not only TAMs, but also circulating monocytes and bone marrow (BM) myeloid progenitors are functionally reprogrammed by tumor-derived factors even before their recruitment in the TME.
2. Radioactive iodide (I131)(RAI) is a very effective therapy for patients with TC, but is less effective in patients with advanced, metastatic tumors. We hypothesize that by exposing tumor antigens to the immune system, RAI might induce immunogenic effects at the level of the TME with reprogramming of both TAMs present in the TME and circulating monocytes, towards a tumor suppressive phenotype. This may further potentiate the effects of RAI. In addition this could be explored in the future as a basis for immunotherapy for tumors that are refractory to conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

* Group 1:

Subject is newly diagnosed with TC, therapy-naive and is planned to receive conventional treatment by surgery followed by RAI; no evidence of local or distant metastases

* Group 2:

Subject has TC with evidence of distant metastases (either newly diagnosed or therapy-naive or patients with persistent or recurrent disease); at least 4 months since the previous treatment with RAI if applicable

* Group 3:

Subject is diagnosed with MNG, is euthyroid, and is planned to undergo surgery - Group 4: Subject is diagnosed with MNG, is euthyroid, and is planned to receive RAI treatment

- Group 5: Healthy individuals who are euthyroid and have no evidence of thyroid disease

Exclusion Criteria:

* Mentally incompetent
* Pregnant, trying to become pregnant or breastfeeding
* Known inflammatory or infectious diseases or an immunosuppressive status
* Using medication interfering with the immune system
* Reduced platelet counts or other conditions associated with an increased risk of bleeding
* Severe comorbidities: other active malignancy (except for basal cell carcinoma)
* Serious psychiatric pathology
* A self-reported alcohol consumption of >21 units per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
Transcriptional reprogramming of myeloid cells | baseline
  RNAseq
Epigenetic reprogramming of myeloid cells | baseline
  ATAC-seq
Functional reprogramming of myeloid cells | baseline
  Cytokine response

SECONDARY OUTCOMES:
Metabolites | baseline
  Presence and level metabolites
Change of reprogramming after RAI treatment | baseline and 7 days after RAI treatment
  RNAseq

CONTACTS AND LOCATIONS:
Overall Officials: Romana T Netea-Maier, Principal Investigator — Endocrinologist
Locations (1):
- Radboudumc, Nijmegen, Netherlands